CLINICAL TRIAL: NCT00397930
Title: Yoga for Persistent Sleep Disturbance in Cancer Survivors
Brief Title: Yoga in Treating Sleep Disturbance in Cancer Survivors
Acronym: YOCAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gary Morrow (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, Gary Morrow, Director, URCC NCORP Research Base, University of Rochester NCORP Research Base
Organization: University of Rochester (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000515123; U10CA037420 (NIH); URCC U3905 (Other: University of Rochester); URCC-04-01 (Other: NCI/DCP)
Record Dates: First submitted 2006-11-09; First posted 2006-11-10 (Estimated); Results first posted 2015-03-17 (Estimated); Last update posted 2017-02-20 (Actual); Status verified 2017-01

CONDITIONS: Fatigue; Cancer; Sleep Disorders
Keywords: cancer-related sleep disturbance; fatigue; sleep disorders
MeSH Terms: conditions — Fatigue; Neoplasms; Sleep Wake Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Yoga Intervention (YOCAS) (Experimental): Standardized Yoga for Cancer Survivors (YOCAS)
  Interventions: Procedure: Yoga Intervention (YOCAS)
- Standard Care Control Condition (Experimental): Standard follow-up care provided by their treating oncologists as appropriate for individual diagnoses.
  Interventions: Procedure: Standard Care Control Condition

INTERVENTIONS:
Procedure: Standard Care Control Condition — Cancer survivors assigned to this condition continued with the standard follow-up care provided by their treating oncologists as appropriate for individual diagnoses. Participants in the control condition were offered the 4-week YOCAS program gratis after completing all study requirements.
  Arms: Standard Care Control Condition
Procedure: Yoga Intervention (YOCAS) — The Yoga for Cancer Survivors (YOCAS) intervention uses two forms of yoga: Gentle Hatha yoga and Restorative yoga. The YOCAS sessions are standardized, and each session includes physical alignment postures, breathing and mindfulness exercises. The intervention is delivered in an instructor taught, group format, twice a week for 75 minutes each time over 4 weeks for a total of eight sessions of yoga. All sessions were taught in community-based sites (eg. yoga studios, community centers, community oncology practices) with an average group size of 12 (range, 10-15) in the late afternoon or evening after 4pm.
  Arms: Yoga Intervention (YOCAS)

SUMMARY:
RATIONALE: Yoga may help improve sleep, fatigue, and quality of life in cancer survivors.

PURPOSE: This phase II trial is studying how well yoga works in treating sleep disturbance in cancer survivors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of Hatha yoga in improving sleep quality in cancer survivors experiencing persistent sleep disturbance.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to gender and sleep disturbance rating reported on the eligibility assessment questionnaire (≤ 5 vs > 5). Patients are randomized to 1 of 2 arms.

* Arm I: Patients receive standard care for 6 weeks. Patients may switch to the yoga intervention immediately after study completion.
* Arm II:Patients receive standard care for 2 weeks, followed by two 75-minute sessions of Hatha yoga per week for 4 weeks.

PROJECTED ACCRUAL: A total of 400 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of any type of cancer
* More than 1 primary cancer allowed
* Has undergone and completed all forms of standard treatment (surgery, chemotherapy, radiation therapy) within the past 2 to 24 months
* Patients can be on hormones such as Tamoxifen, or monoclonal antibodies like Herceptin
* Persistent sleep disturbance, as indicated by a response of ≥ 3 when asked to rate their sleep on an 11-point scale (0 is equivalent to no sleep disturbance and 10 is the worst possible sleep disturbance)
* Able to read English
* 21 years of age or older

Exclusion Criteria:

* No prior or concurrent regular (≥ 1 day/week) participation in yoga classes or maintain regular personal practice of any form of yoga within the past 3 months
* No diagnosis of sleep apnea
* No concurrent cancer therapy with the exception of hormonal therapy (e.g., tamoxifen citrate) or monoclonal antibodies (e.g., trastuzumab [Herceptin®])
* No metastatic cancer

Ages: 21 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Actual)
Dates: Start 2006-10; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen M. Mustian, PhD, Principal Investigator — University of Rochester
Locations (11):
- United States (11):
  - CCOP - Central Illinois, Decatur, Illinois
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Hematology-Oncology Associates of Central New York, East Syracuse, New York
  - CCOP - Southeast Cancer Control Consortium, Goldsboro, North Carolina
  - CCOP - Columbus, Columbus, Ohio
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Northwest, Tacoma, Washington

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Messer S, Oeser A, Wagner C, Wender A, Cryns N, Scherer RW, Mishra SI, Monsef I, Holtkamp U, Andreas M, Brockelmann PJ, Ernst M, Skoetz N. Yoga for fatigue in people with cancer. Cochrane Database Syst Rev. 2025 May 27;5(5):CD015520. doi: 10.1002/14651858.CD015520. PMID 40421669
- [Derived] Arana-Chicas E, Lin PJ, Gada U, Sun H, Chakrabarti A, Mattick LJ, Rieth K, Chay CH, Ruzich J, Esparaz BT, Cupertino AP, Altman BJ, Vertino PM, Mohile SG, Mustian KM. The effect of YOCAS(c)(R) yoga on cancer-related fatigue and quality of life in older (60+) vs. younger (</= 59) cancer survivors: Secondary analysis of a nationwide, multicenter, phase 3 randomized controlled trial. J Geriatr Oncol. 2024 Nov;15(8):102076. doi: 10.1016/j.jgo.2024.102076. Epub 2024 Oct 4. PMID 39368335
- [Derived] Lin PJ, Kleckner IR, Loh KP, Inglis JE, Peppone LJ, Janelsins MC, Kamen CS, Heckler CE, Culakova E, Pigeon WR, Reddy PS, Messino MJ, Gaur R, Mustian KM. Influence of Yoga on Cancer-Related Fatigue and on Mediational Relationships Between Changes in Sleep and Cancer-Related Fatigue: A Nationwide, Multicenter Randomized Controlled Trial of Yoga in Cancer Survivors. Integr Cancer Ther. 2019 Jan-Dec;18:1534735419855134. doi: 10.1177/1534735419855134. PMID 31165647
- [Derived] Mustian KM, Sprod LK, Janelsins M, Peppone LJ, Palesh OG, Chandwani K, Reddy PS, Melnik MK, Heckler C, Morrow GR. Multicenter, randomized controlled trial of yoga for sleep quality among cancer survivors. J Clin Oncol. 2013 Sep 10;31(26):3233-41. doi: 10.1200/JCO.2012.43.7707. Epub 2013 Aug 12. PMID 23940231
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — https://www.cancer.gov/publications/pdq

RESULTS

PARTICIPANT FLOW:
Groups:
- Yoga Intervention (YOCAS): The yoga intervention used the standardized Yoga for Cancer Survivors (YOCAS) program, designed by researchers at the University of Rochester Medical Center. All sessions were taught in community-based sites (eg. yoga studios, community centers, community oncology practices) with an average group size of 12 (range, 10-15) in the late afternoon or evening after 4pm.
  fatigue assessment and management
  management of therapy complications
  quality-of-life assessment
  sleep disorder therapy
  yoga therapy
- Standard Care Control Condition: The control condition used a standard care format. Cancer survivors assigned to this condition continued with the standard follow-up care provided by their treating oncologists as appropriate for individual diagnoses. Participants in the control condition were offered the 4-week YOCAS program gratis after completing all study requirements.
  fatigue assessment and management
  management of therapy complications
  quality-of-life assessment
Period: Overall Study
Arm/Group | Yoga Intervention (YOCAS) | Standard Care Control Condition
Started | 206 | 204
Completed | 168 | 153
Not Completed | 38 | 51
Not completed — Personal reasons | 14 | 8
Not completed — Other medical | 9 | 4
Not completed — Unknown reasons | 9 | 14
Not completed — Noncompliant | 3 | 2
Not completed — Too time-consuming | 2 | 9
Not completed — Started own yoga program | 1 | 1
Not completed — Did not want to be in control group | 0 | 1
Not completed — Withdrawal by Subject | 0 | 8
Not completed — Missing data | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Yoga Intervention (YOCAS) | Standard Care Control Condition | Total
Number analyzed (Participants) | 206 | 204 | 410
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 54.3 (11.05) | 54 (9.57) | 54.1 (10.33)
Gender [Count of Participants; unit: Participants]
  Female | 197 | 196 | 393
  Male | 9 | 8 | 17
Race/Ethnicity, Customized [Number; unit: participants]
  White | 197 | 186 | 383
  African American | 8 | 16 | 24
  Other | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 206 | 204 | 410
Currently employed [Number; unit: participants]
  Yes | 168 | 155 | 323
  No | 38 | 49 | 87
Marital status [Number; unit: participants]
  Married or long-term committed relationship | 145 | 143 | 288
  Divorced or separated | 28 | 32 | 60
  Single | 18 | 17 | 35
  Widowed | 6 | 12 | 18
  Unknown | 9 | 0 | 9
Education [Number; unit: participants]
  Completed 4 years of college or more | 96 | 93 | 189
  Completed < 4 years of college | 72 | 69 | 141
  High school graduate | 33 | 36 | 69
  Less than a high school graduate | 2 | 1 | 3
  Unknown | 3 | 5 | 8
Cancer type [Number; unit: participants]
  Breast | 152 | 157 | 309
  Hematologic | 16 | 14 | 30
  Gynecologic | 11 | 8 | 19
  Alimentary | 7 | 17 | 24
  Other | 20 | 8 | 28
Cancer stage [Number; unit: participants]
  0 | 11 | 10 | 21
  I | 66 | 79 | 145
  II | 71 | 66 | 137
  III | 32 | 32 | 64
  IV | 7 | 4 | 11
  Unknown | 19 | 13 | 32
Previous treatment - Surgery [Number; unit: participants]
  Yes | 183 | 181 | 364
  No | 23 | 23 | 46
Previous Treatment - Chemotherapy [Number; unit: participants]
  Yes | 145 | 139 | 284
  No | 61 | 65 | 126
Previous Treatment - Radiation therapy [Number; unit: participants]
  Yes | 137 | 129 | 266
  No | 69 | 75 | 144
Previous Treatment - Hormone treatment [Number; unit: participants]
  Yes | 13 | 15 | 28
  No | 193 | 189 | 382
Current hormone therapy [Number; unit: participants]
  Yes | 99 | 107 | 206
  Unknown | 107 | 97 | 204
Time since first treatment for cancer [Mean (Standard Deviation); unit: months] | 14.9 (7.18) | 17.7 (23.00) | 16.3 (17.00)
Karnofsky performance status [Mean (Standard Deviation); unit: Karnofsky performance scale] — The Karnofsky Performance Scale (KPS) Index allows patients to be classified as to their functional impairment. Essentially as used in oncology, the KPS is a measure of time to death. A higher score is favorable. There are 3 general categories which are broken down into 11 specific criteria. Scale range is from 0 (Dead) to 100 (Normal, no complaints, no evidence of disease). The scale increases in units of 10.
  Karnofsky performance scale | 86.9 (33.15) | 87.8 (32.00) | 87.4 (32.6)
Exercise stage of change [Number; unit: participants]
  Not exercising and do not intend to in next 6 mo | 8 | 10 | 18
  Not exercising but intend to in next 6 mo | 43 | 38 | 81
  Not exercising but intend to begin in next 30 days | 45 | 50 | 95
  Exercising and have been for less than 6 months | 44 | 43 | 87
  Exercising and have been for more than 6 months | 62 | 58 | 120
  Unknown | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Mean Post-Pre Change for the Pittsburgh Sleep Quality Inventory (PSQI)
Description: Pittsburgh Sleep Quality Index: Measures sleep disturbance and usual sleep habits during the prior month only using seven clinically derived domains of sleep difficulties: sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medications, and daytime dysfunction. Global PSQI is a summary of the seven domains. Each Domain is scored from 0 to 3, therefore PSQI has a range of 0 (better) to 21 (worse). Interpretation of the PSQI is that a score less than 5 is associated with good sleep quality and a score of 5 or greater is associated with poor sleep quality.
  PSQI was calculated at both pre- and post-intervention for both arms. Pre-intervention PSQI was recorded during the week immediately before commencing the 4-week intervention. Post-intervention PSQI was recorded during the week immediately following the intervention. Mean post-pre change was calculated for both arms.
Time Frame: 2-24 months after surgery, chemotherapy, and/or radiation therapy
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Yoga Intervention (YOCAS) | Standard Care Control Condition
Number analyzed (Participants) | 168 | 153
units on a scale | -1.96 (0.25) | -1.07 (0.23)
Statistical Analysis 1: Comparison: Yoga Intervention (YOCAS) vs Standard Care Control Condition; H0: There is no statistically significant difference in global sleep quality between post-treatment cancer survivors under the standardized yoga intervention and control protocol at the 0.05 two-sided significance level. Ha: There is a statistically significant difference in global sleep quality between post-treatment cancer survivors under the standardized yoga intervention and control protocol at the 0.05 two-sided significance level; Test type: Superiority or Other; p = 0.009, ANCOVA — Between-group differences are expressed as differences in mean Post-Pre change for the global sleep quality PSQI score; ANCOVA with post-intervention PSQI score as the outcome, with Group as the factor, and pre-intervention PSQI score as the covariate; Mean Difference (Final Values) = -0.79, Standard Error of Mean 0.30 — The negative estimated value indicates that the mean Post-Pre change for the YOCAS group was less than that of the Control group

ADVERSE EVENTS:
Arm/Group | Yoga Intervention (YOCAS) | Standard Care Control Condition
Serious Adverse Events (participants affected / at risk) | 1/206 | 1/204
Other Adverse Events (participants affected / at risk) | 0/206 | 0/204
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Yoga Intervention (YOCAS) (N=206) | Standard Care Control Condition (N=204)
Death (General disorders) | 1 | 0 — hosp d/t abd pain
Death (Metabolism and nutrition disorders) | 0 | 1 — Dehydration

LIMITATIONS AND CAVEATS:
The study did not account for components such as time or attention, as this would have required the use of a placebo yoga intervention for the YOCAS program. The results are not generalizable for all yoga types, nor for all socioeconomic backgrounds.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No